CLINICAL TRIAL: NCT01986361
Title: A Single-Dose, Randomized, Double-Blind, Placebo-Controlled Onset-of-Action Study Utilizing the Double-Stopwatch Method
Brief Title: Placebo-Controlled Onset-of-Action Study of Flurbiprofen Utilizing the Double-Stopwatch Method
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-STR-01
Record Dates: First submitted 2013-10-22; First posted 2013-11-18 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Acute Pharyngitis; Sore Throat
Keywords: Pharyngitis; Sore Throat; acute upper respiratory tract infection (URTI)
MeSH Terms: conditions — Pharyngitis | interventions — Flurbiprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- flurbiprofen 8.75 mg lozenge (Experimental): A single flurbiprofen lozenge is sucked until fully dissolved.
  Interventions: Drug: flurbiprofen
- Placebo lozenge (Placebo Comparator): A single placebo lozenge is sucked until fully dissolved.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: flurbiprofen — A single flurbiprofen 8.75 mg lozenge which also contains 1 mg of menthol in its vehicle base for flavour and taste purposes (blinding). Lozenge is sucked until dissolved, and not chewed, bit or swallowed.
  Arms: flurbiprofen 8.75 mg lozenge
Drug: placebo — A single placebo lozenge which also contains 1 mg of menthol in its vehicle base for flavour and taste purposes (blinding). Lozenge is sucked until dissolved, and not chewed, bit or swallowed.
  Arms: Placebo lozenge

SUMMARY:
The study's purpose is to demonstrate the onset of action, i.e., time to meaningful pain relief in patients with pharyngitis, of flurbiprofen 8.75 mg lozenge using the Double-Stopwatch Method (DSW).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: pharyngitis confirmed by a Tonsillo-Pharyngitis Assessment ≥ 5
* Complaint of sore throat with an onset ≤ 4 days prior to randomization
* Have at least one symptom of upper respiratory tract infection (URTI) on the URTI Questionnaire (e.g., sore throat, runny nose, cough, fever)
* Have moderate or severe sore throat pain on the Throat Pain Scale
* Have a baseline Sore Throat Scale (STS) ≥ 6
* If the patient is a female of childbearing potential, she has been using effective contraception since the last date of menses and is not breast-feeding or lactating. She is also willing to take adequate contraceptive precautions through 24 hours after the completion of the study.
* If the patient is a female of childbearing potential, the patient must have a negative urine pregnancy test (UPT) result (indicating "not pregnant") obtained on the day of scheduled randomization, prior to the designated time of randomization
* The patient is willing to remain at the study centre for 3 hours after receiving the dose of study medication
* During the 3-hour evaluation of the study medication lozenge at the site, the patient is willing to take "nothing by mouth" (e.g., no smoking, food, candy, lozenges, chewing gum, liquids).

Exclusion Criteria:

* Known allergy and/or hypersensitivity to aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), or any other inactive ingredients such as honey, lemon flavor, menthol, or sucrose.
* History of an upper gastrointestinal ulcer within the past 60 days, current clinically significant upper gastrointestinal complaints, or current regular use (≥ 3 times in the previous week) of any medication for upper gastrointestinal symptoms, including antacids, H2 blockers, proton pump inhibitors or sucralfate
* History of any hepatic disease or renal dysfunction
* Other severe acute or chronic medical condition that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
* History of chronic analgesic use (≥ 3 times per week over the prior 4 weeks)
* Use of an antibiotic for an acute disease within the previous 24 hours before randomization. (Chronic antibiotic use, such as for acne, is acceptable.) Use of any quinolone antibiotic such as ciprofloxacin or nalidixic acid within the past week or concurrently is specifically prohibited.
* Use of mifepristone in the 12 days prior to the screening visit
* Use of inhaled therapy (e.g., inhaled steroids or β-agonists, such as Ventolin) on an acute basis for disease exacerbation in the week prior to the screening visit
* Use of any immediate release analgesic within 4 hours preceding administration of the study medication.
* Use of any sustained release analgesic within 12 hours preceding administration of the study medication.
* Use of any "cold medication" (i.e. decongestants, antihistamines, expectorants, antitussives) within 4 hours preceding administration of the dose of study medication.
* Use of any throat lozenge, throat spray, cough drop, or menthol-containing product within 2 hours preceding administration of the study medication
* Consumption of any caffeine-containing beverage (e.g., coffee, tea, hot chocolate, caffeinated soft drinks) within 5 minutes preceding administration of the study medication.
* Any evidence of mouth-breathing (which could worsen sore throat pain).
* Coughing that causes throat discomfort or any active physical disease (such as bronchopneumonia) which could compromise respiratory function and worsen a sore throat
* Unable in the opinion of the Investigator to comply fully with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Shea, BS, Study Director — Reckitt Benckiser Inc.
Locations (1):
- University of Connecticut - Student Health Services, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Schachtel B, Shephard A, Schachtel E, Lorton MB, Shea T, Aspley S. Qualities of Sore Throat Index (QuaSTI): measuring descriptors of sore throat in a randomized, placebo-controlled trial. Pain Manag. 2018 Mar;8(2):85-94. doi: 10.2217/pmt-2017-0041. Epub 2018 Jan 30. PMID 29381110

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 133 patients were screened and 122 enrolled. Participants were randomly assigned in a 5:1 ratio to receive either an 8.75 mg flurbiprofen lozenge or a vehicle lozenge (placebo).
Period: Overall Study
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Started | 101 | 21
Completed | 101 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge | Total
Number analyzed (Participants) | 101 | 21 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (2.02) | 19.6 (1.36) | 19.5 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 13 | 71
  Male | 43 | 8 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Non-Hispanic or Non-Latino | 93 | 19 | 112
Primary Race [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black or African American | 3 | 2 | 5
  Multi-Racial | 2 | 0 | 2
  White | 94 | 19 | 113
Weight [Mean (Standard Deviation); unit: pounds] | 154.09 (31.221) | 154.19 (35.885) | 154.11 (31.913)
Height [Mean (Standard Deviation); unit: inches] | 67.67 (4.187) | 66.90 (3.697) | 67.54 (4.103)
Sore Throat Scale (STS) Score [Mean (Standard Deviation); unit: units on a scale] — The participant was asked to evaluate his/her sore throat when swallowing using a vertical 0-10 Likert scale, where 0=not sore and 10=very sore. The participant was instructed: "Circle the number that shows how sore your throat is now when you swallow."
  units on a scale | 7.4 (0.97) | 7.3 (1.02) | 7.4 (0.98)
Sore Throat Pain Intensity Scale (STPIS) [Mean (Standard Deviation); unit: units on a scale] — The participant was instructed to swallow and: "Place a line on the Sore Throat Scale that best characterizes the severity of your sore throat now:" 0mm=no pain and 100mm=severe pain.
  units on a scale | 73.8 (9.78) | 73.8 (9.64) | 73.8 (9.71)

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates for Time to Meaningful Pain Relief
Description: Time to meaningful pain relief is a patient-reported outcome (PRO) captured as part of the double stopwatch method. Participants depress the second stop watch when they experience what they perceive as meaningful pain relief. Instructions to participants are: "Stop the second stopwatch when the sore throat pain relief is meaningful to you. This does not mean you feel completely better, although you might, but when you feel relief of throat pain that is meaningful to you." Participants who did not have perceived pain relief were censored at 3 hours.
Time Frame: up to 3 hours post dose on Day 1
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
minutes | 42.917 [36.367 to 49.383] | NA [47.567 to NA] — Less than 50% achieved meaningful relief

2. Secondary Outcome: Kaplan-Meier Estimates for Time of First Perceived Pain Relief
Description: Time to first perceived pain relief is a patient-reported outcome (PRO) captured as part of the double stopwatch method. Participants depress the first stop watch when they experience any pain relief, termed "perceived pain relief". Instructions to participants are: "Stop the first stopwatch when you first feel any sore throat pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief of the throat pain you have now." Participants who did not have perceived pain relief were censored at 3 hours.
Time Frame: up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
minutes | 10.867 [7.633 to 14.283] | 19.317 [4.783 to 30.333]

3. Secondary Outcome: Kaplan-Meier Estimates for Time to First Perceived Pain Relief That Is Confirmed By Meaningful Pain Relief
Description: Time to first perceived pain relief on the first stopwatch that was confirmed by meaningful pain relief on the second stopwatch. Participants who had no meaningful pain relief within 3 hours from baseline were censored to 3 hours.
Time Frame: up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
minutes | 13.200 [8.633 to 16.567] | NA [6.633 to NA] — Less than 50% achieved meaningful relief

4. Secondary Outcome: Kaplan-Meier Estimates for Time of First Indication of Sore Throat Relief as Measured By Any Reduction in the Sore Throat Scale (STS)
Description: Time to first indication of sore throat relief, defined as any reduction or decrease in STS observed during the 3 hours post dose. Participants who did not have any reduction in STS from baseline within 3 hours were censored to 3 hours.
  The participant was asked to evaluate his/her sore throat when swallowing using a vertical 0-10 Likert scale, where 0=not sore and 10=very sore. The participant was instructed: "Circle the number that shows how sore your throat is now when you swallow." The STS was obtained at baseline, every 5 minutes after treatment during the first hour and every 10 minutes during the second and third hours.
Time Frame: up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
minutes | 15.000 [10.000 to 15.000] | 20.000 [5.000 to 30.000]

5. Secondary Outcome: Kaplan-Meier Estimates for Time of First Perceived Pain Reduction on the Sore Throat Scale (STS) Which is Followed by ≥ 20% Pain Reduction on the Sore Throat Pain Intensity Scale (STPIS)
Description: Time to pain reduction on the STS (defined as any reduction or decrease observed during the 3 hours post dose) for participants whose improvement was confirmed by a >=20% reduction in pain on the STPIS.
  STS: The participant was asked to evaluate his/her sore throat when swallowing using a vertical 0-10 Likert scale, where 0=not sore and 10=very sore. The participant was instructed: "Circle the number that shows how sore your throat is now when you swallow." The STS was obtained at baseline, every 5 minutes after treatment during the first hour and every 10 minutes during the second and third hours.
  STPIS: The participant was instructed to swallow and: "Place a line on the Sore Throat Scale that best characterizes the severity of your sore throat now:" 0mm=no pain and 100mm=severe pain. The STPIS was obtained at baseline, after the participant depressed the second stopwatch, and at 1, 2, and 3 hours postdose.
Time Frame: Baseline (Day 1, pre-dose), up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
minutes | 15.000 [10.000 to 20.000] | NA [10.000 to NA] — Less than 50% achieved confirmed relief

6. Secondary Outcome: Change From Baseline at Individual Timepoints in Sore Throat Scale (STS)
Description: The participant was asked to evaluate his/her sore throat when swallowing using a vertical 0-10 Likert scale, where 0=not sore and 10=very sore. The participant was instructed: "Circle the number that shows how sore your throat is now when you swallow." The STS was obtained at baseline, every 5 minutes after treatment during the first hour and every 10 minutes during the second and third hours.
Time Frame: Baseline (Day 1, pre-dose), up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
units on a scale
  Minute 5 | -0.4 (0.90) | -0.4 (0.67)
  Minute 10 | -0.7 (1.14) | -0.6 (0.98)
  Minute 15 | -0.9 (1.26) | -0.6 (0.87)
  Minute 20 | -1.0 (1.30) | -0.6 (0.74)
  Minute 25 | -1.3 (1.34) | -0.7 (0.90)
  Minute 30 | -1.6 (1.41) | -1.0 (1.12)
  Minute 35 | -1.8 (1.52) | -1.0 (1.20)
  Minute 40 | -2.0 (1.50) | -1.1 (1.34)
  Minute 45 | -2.2 (1.54) | -1.2 (1.36)
  Minute 50 | -2.3 (1.59) | -1.3 (1.52)
  Minute 55 | -2.4 (1.64) | -1.1 (1.49)
  Minute 60 | -2.5 (1.69) | -1.1 (1.65)
  Minute 70 | -2.6 (1.74) | -1.2 (1.72)
  Minute 80 | -2.7 (1.85) | -1.1 (1.61)
  Minute 90 | -2.7 (1.86) | -1.0 (1.77)
  Minute 100 | -2.7 (1.87) | -1.0 (1.72)
  Minute 110 | -2.7 (1.85) | -1.0 (1.83)
  Minute 120 | -2.7 (1.91) | -1.0 (1.94)
  Minute 130 | -2.6 (1.86) | -1.0 (1.83)
  Minute 140 | -2.6 (1.95) | -0.9 (1.82)
  Minute 150 | -2.5 (1.99) | -0.8 (1.97)
  Minute 160 | -2.4 (2.01) | -0.9 (2.06)
  Minute 170 | -2.3 (2.06) | -0.8 (2.23)
  Minute 180 | -2.3 (2.05) | -0.8 (2.06)

7. Secondary Outcome: Percentage of Participants With Meaningful Pain Relief
Description: Defined as the percentage of participants who pressed the second stopwatch during the 3 hour evaluation period.
Time Frame: up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
percentage of participants | 78.2 [70.2 to 86.3] | 47.6 [26.3 to 69.0]

8. Secondary Outcome: Percentage of Participants With Perceived Pain Relief
Description: Defined as the percentage of participants who pressed the first stopwatch during the 3 hour evaluation period.
Time Frame: up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
percentage of participants | 97.0 [93.7 to 100.0] | 76.2 [58.0 to 94.4]

9. Secondary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Scale (STS) Over the 3 Hours Post-baseline (STS SPID3)
Description: The participant was asked to evaluate his/her sore throat when swallowing using a vertical 0-10 Likert scale, where 0=not sore and 10=very sore. The participant was instructed: "Circle the number that shows how sore your throat is now when you swallow." STS was obtained at baseline, every 5 minutes after treatment during the first hour and every 10 minutes during the second and third hours, for a total of 24 post-dose measurements.
  The time-weighted SPID combines relief magnitude (PID = change from baseline) as weighted by duration interval between ratings. SPID3 refers to measurements taken up to 3 hours post-baseline, and has a full range of -1332 (complete pain relief within 5 minutes of dosing that lasts for 3 hours) to 468 (drug escalates level of pain to a score of 10 and the pain stays at that level for 3 hours) using the mean baseline STS value 7.4 for this study.
Time Frame: Baseline (Day 1, pre-dose), up to 3 hours post dose on Day 1
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 21
units on a scale | -403.9 [-457.3 to -350.5] | -166.4 [-286.8 to -46.0]

ADVERSE EVENTS:
Time Frame: up to 20 hours post dose
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/21
Other Adverse Events (participants affected / at risk) | 10/101 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flurbiprofen 8.75 mg Lozenge (N=101) | Placebo Lozenge (N=21)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.